CLINICAL TRIAL: NCT05906017
Title: Open Versus Robotic-assisted Ventral Hernia Repair, Short and Long-term Outcome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS-MT Kir-2-2023
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Abdominal Hernia
Keywords: Da Vinci; Robot; Umbilical hernia; Ventral hernia; Epigastric hernia; Hernia repair; Laparotomy
MeSH Terms: conditions — Hernia, Abdominal; Hernia, Umbilical; Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open repair (Active Comparator): Open ventral hernia repair
  Interventions: Procedure: Open Hernia surgery
- Robotic-assisted repair (Experimental): Robotic-assisted ventral hernia repair
  Interventions: Procedure: Robotic Hernia surgery

INTERVENTIONS:
Procedure: Open Hernia surgery — midline ventral hernia repair - open
  Arms: Open repair
Procedure: Robotic Hernia surgery — midline ventral hernia repair - robotic
  Arms: Robotic-assisted repair

SUMMARY:
In this randomized clinical trial, the investigators will compare the conventional open repair for hernia in the anterior abdominal wall with the robotic-assisted approach. 60 patients with midline abdominal wall defects will be randomized to either open or robotic-assisted surgery. The investigators will examine short and long-term complications through follow-up with clinical assessment as well as patient-reported outcome measures including pain, cosmetic appearance, and overall patient satisfaction. Furthermore, the investigators will study the difference in surgical stress response between the two methods measured from a variety of different biomarkers before and after the operation. A cost-effective analysis will be conducted for the robotic and open procedure.

DETAILED DESCRIPTION:
Ventral hernias occur in up to 25% of the population. They are diverse in severity ranging from small umbilical hernias to large abdominal wall defects that may result in loss of domain. Approximately one-third are incisional hernias. Incisional hernias are usually more complex due to complications from previous surgery. The procedure may be complicated as a result of intraabdominal bowel adhesions and adhesions within the hernial sac. These factors cause discomfort and may complicate the repair. Ventral hernias may be repaired either through a minimally invasive laparoscopic procedure or an open approach. The laparoscopic repair was introduced in the 1990s and in 2003 the first robotic-assisted procedure was described in a porcine model. In 2012 the first series of robotic repairs were reported in humans. Due to the superior flexibility of the robotic instruments, there is a substantial interest in harnessing the advantages of the robotic platform. Because robotic repair differs in several technical aspects from the open approach, it is important to determine whether the short and long-term results differ between the two procedures. Furthermore, it remains unresolved whether the robotic procedure is able to provide comparable outcomes to the open repair when assessed for quality-of-life outcome measures. These questions are important to address in order to determine the most appropriate surgical options for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* ASA 1-3
* Clinical and radiologic diagnosis of midline ventral hernia
* Eligible to surgery according to a preoperative anaesthetic assessment
* Informed consent
* Able to understand written and oral Danish language

Exclusion Criteria:

* Incarcerated ventral hernia requiring emergency surgery
* Pregnancy
* Patients with chronic pain due to arthritis, migraine or other illness requiring regular intake of analgesics (paracetamol, NSAID, opiates etc).
* Current cancer diagnosis
* History of psychiatric or addictive disorder that prevents the patient from participating in the trial
* Co-existing inflammatory disease
* Co-existing immunological disease that requires medication of any kind
* BMI >40 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Length of stay (LOS) | Up until 3 months
  The primary outcome measure will be assessed by reviewing the electronic patient journal system. The day of the procedure will be recorded as day 0

SECONDARY OUTCOMES:
Operating time | Time from first incision to wound closure
  Measured in minutes
Change in Surgical stress response (CRP) | measured at baseline preoperatively, 30 minutes after extubation, 120 minutes after extubation and on day 1 and 3.
  The degree of systemic inflammatory response expressed by C- reactive protein in serum
Hernia defect size | Measured preoperatively
  Hernia defect size measured in mm either on CT scan or intraoperative.
Intraoperative need of blood transfusion | From first incision until last suture has been placed
  The amount of blood transfused during surgery measured in mL
Change in surgical stress response (Interleukins) | Measured at baseline preoperatively and up until 120 minutes after extubation on day 1 and 3.
  The degree of systemic inflammatory response expressed by cytokine levels in serum. All measurements will consist of weight/volume ratio (eg. CRP mg/L and IL-6 pg/mL)
Treatment cost | From inclusion until 6 months postoperatively
  Cost analysis of the two types of treatment
Change in satisfaction and quality of life | [Time Frame: From inclusion until 6 months after operation.]
  Satisfaction and quality of life were measured preoperatively at the outpatient clinic using the "abdominal hernia questionnaire" (AHQ) translated into Danish. The AHQ has 4 possible answers (All of the time, Most of the time, Some of the time, None the time OR Strongly disagree, Somewhat disagree, Somewhat agree, Strongly agree OR Very unsatisfied, Somewhat dissatisfied, Somewhat satisfied, Very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Festersen Nielsen, Study Director — Hospital of Southern Denmark - Aabenraa
Locations (1):
- Sygehus Sønderjylland, Aabenraa, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No